CLINICAL TRIAL: NCT06814496
Title: RAdiation comBined With BIspecific T-Cell Engager in DLL3 Expressing Tumors (RABBIT) Study: A Phase I/II Study of AMG757 / Tarlatamab and Concurrent Radiation Therapy in Tumors With High Prevalence of DLL3
Brief Title: Radiation Combined With BIspecific T-Cell Engager in DLL3 Expressing Tumors
Acronym: RABBIT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005401; 20247128 (Other Grant/Funding Number: Amgen)
Record Dates: First submitted 2025-01-29; First posted 2025-02-07 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Melanoma; Medullary Thyroid Cancer; Sinonasal Undifferentiated Carcinoma; Esthesioneuroblastoma; Bladder Cancer; Testicular Cancer; Glioblastoma Multiforme; Cervical Cancer; Large Cell Neuroendocrine Carcinoma of the Lung; Non Small Cell Lung Cancer; Merkel Cell Carcinoma
Keywords: DLL3 Expressing tumors
MeSH Terms: conditions — Melanoma; Carcinoma, Medullary; Sinonasal undifferentiated carcinoma; Esthesioneuroblastoma, Olfactory; Urinary Bladder Neoplasms; Testicular Neoplasms; Glioblastoma; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Merkel Cell

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled on the Concurrent Main Cohort (tarlatamab with concurrent radiation therapy to extracranial sites; N=20-24 extracranial RT site with a minimum of 10 thoracic patients). If the safety endpoint is met, enrollment will expand to the Concurrent Cranial Cohort (tarlatamab with concurrent radiation therapy to cranial sites; N=6-10 cranial RT sites).
  If the concurrent safety endpoint is not met, then the study will proceed to the de-escalation phase, where patients will be enrolled on the Sequential Cohort (sequential tarlatamab and radiation therapy; N=20 cranial and extracranial RT sites).
  If the sequential safety endpoint is not met, then the study will proceed to another de-escalation phase, where patients will be enrolled on the Tarlatamab Monotherapy Cohort (N=10 enriched for non-tumors not of SCLC tumorshistology and allowing for patients without amenable RT sites).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Concurrent Main Cohort (Experimental): Patients enrolled to this cohort will receive tarlatamab with concurrent radiation therapy (RT) to extracranial sites (n=20-24 extracranial RT with a minimum of 10 thoracic patients). Patients will receive tarlatamab at a step-up dose of 1 mg on Cycle 1 Day 1 and then 10 mg on cycle 1 Day 8 and Cycle 1 Day 15 and every 2 weeks thereafter (on days 1 and 15 of each cycle) until radiographic progression or disease progression or 24 months, whichever is earlier. Patients will receive concurrent RT to extracranial sites as per standard of care starting as early as Cycle 1 Day 16 and as late as Cycle 2 Day 28, assuming there is no ongoing cytokine release syndrome (CRS) or immune-effector cell-associated neurotoxicity Syndrome (ICANS).
  Interventions: Drug: Tarlatamab; Radiation: Concurrent Radiation Therapy
- Concurrent Cranial Cohort (Experimental): If the safety endpoint in the Concurrent Main Cohort is met, enrollment will expand to the Concurrent Cranial Cohort. 6-10 patients will receive tarlatamab with concurrent radiation therapy to cranial sites as described in the Concurrent Main Cohort.
  Interventions: Drug: Tarlatamab; Radiation: Concurrent Radiation Therapy
- Sequential radiation therapy cohort (Experimental): If the concurrent main cohort safety endpoint is not met, then the study will proceed to de-escalation, where 20 patients will be enrolled on the sequential radiation therapy cohort. In this cohort patients will receive sequential tarlatamab and RT to cranial and extracranial RT sites. Standard of care RT can occur prior to Cycle 1 Day 1(if radiation treatment is completed <7 days prior to the start of tarlatamab) or be interdigitated with tarlatamab with a 7-day washout between RT and infusion, with RT to begin as early as Cycle 1 Day 22 and as late as cycle 2 Day 28, assuming no ongoing CRS/ICANS.
  Interventions: Drug: Tarlatamab; Radiation: Sequential Radiation therapy
- Tarlatamab Monotherapy Cohort (Experimental): If the sequential safety endpoint is not met, then the study will proceed to another de-escalation phase, where 10 patients will receive tarlatamab alone.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered at a step-up dose of 1mg on Cycle 1 Day 1 and then 10 mg on Cycle 1 Day 8 and Cycle 1 Day 15 and every 2 weeks thereafter. For cycle 2 onwards, tarlatamab infusion will occur every 2 weeks on days 1 and 15 of each cycle.
Radiation: Concurrent Radiation Therapy — Standard of care RT can begin as early as Cycle 1 Day 16 and as late as Cycle 2 Day 28, assuming there is no ongoing CRS (extracranial)/ICANS (cranial).
  Arms: Concurrent Cranial Cohort; Concurrent Main Cohort
Radiation: Sequential Radiation therapy — Standard of care radiation therapy can occur prior to Cycle 1 Day 1 (if radiation treatment is completed <7 days prior to the start of tarlatamab) or be interdigitated with tarlatamab with a 7-day washout between RT and infusion, with RT to begin as early as Cycle 1 Day 22 and as late as cycle 2 Day 28, assuming no ongoing CRS (extracranial)/ICANS (cranial).
  Arms: Sequential radiation therapy cohort

SUMMARY:
Phase I study to examine safety of the addition of concurrent tarlatamab with standard palliative and consolidative RT regimens , with a main cohort of N=20-24 patients with extracranial anatomic radiation sites.

I) After lead in of 10 patients demonstrating safety of treatment, allow for expansion to cranial sites of disease (N=6-10) with continued enrollment in main cohort II) If toxicity criteria is not met in concurrent RT tarlatamab cohort, we will continue with sequential RT, either A) delivered within 7 days prior to cycle 1 day 1, or B) delivered during cycle 1 -2 but with pre- and post-RT washout of 7 days with no drug during RT, to examine safety in a temporally spaced setting.

III) If sequential tarlatamab and radiation is not deemed safe, we would allow for continued enrollment to assess efficacy of drug sans radiation treatment, enriching for tumors not of small cell lung cancer histology and allowing for patients without sites amenable to RT.

A nested phase II study will attempt to assess for ORR and safety of study intervention amongst tumors not of small cell lung cancer histology.

DETAILED DESCRIPTION:
This is a Phase I, Open label, Single Arm, Multi-center Study, with nested Phase II to examine safety of standard palliative and consolidative RT regimens in a main cohort of patients with tumor histologies with high prevalence of DLL3 (N=20-24) with an extracranial site (primary or metastatic) amenable to radiation (not allowing for re-irradiation of the same lesion, with a minimum of 10 thoracic sites. Given the potential toxicity of ICANS with tarlatamab, once deemed safe in the main cohort, we will allow for expansion for treatment of cranial sites amenable to radiation (excluding lesion re-irradiation except for stereotactic radiosurgery / fractionated stereotactic radiosurgery [SRS/fSRS] after prior whole brain RT or prophylactic cranial irradiation [PCI]) with continued enrollment in the main cohort.

Given the need to determine safety of administration of tarlatamb with RT, if safety is not met for concurrent administration in the main cohort, we would discontinue concurrent treatment, and assess safety in a sequential RT and tarlatamab cohort, as temporal de-escalation. If safety is not met in the sequential cohort, treatment with RT will be discontinued and enrollment will continue with tarlatamab monotherapy, not requiring patients having a site amenable to RT and enriching for patients without SCLC.

In the nested phase II, we will assess efficacy of radiation and tarlatamab amongst patients with tumors with high prevalence of DLL3 or those who have positive DLL3 (≥1% per IHC), including but not exclusive to SCLC. This would allow for potential evaluation of safety and response for tumors beyond the DeLLPhi 300/301 studies.

The study population will include patients ≥18 years of age with primary/metastatic sites amenable to external beam radiation treatment refractory solid tumors of:

1. small cell histology
2. high grade / poorly differentiated neuroendocrine histology
3. tumor histologies with high prevalence of DLL3 (≥ 50% prevalence), including but not limited to: melanoma, medullary thyroid cancer, sinonasal undifferentiated carcinoma, esthesioneuroblastoma, bladder cancer, testicular cancer, glioblastoma multiforme, cervical cancer; large cell neuroendocrine tumor of lung, non-small cell lung cancers with mixed neuroendocrine features, and Merkel cell carcinoma OR
4. Patients with DLL3+ tumors (≥1% IHC)

Up to 30 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent/assent prior to initiation of any study specific activities/procedures.
2. Subjects ≥ 18 years of age at the time of signing the informed consent.
3. Histologically or cytologically confirmed relapsed/refractory:

   1. SCLC
   2. Other tumors of small cell histology
   3. High grade / poorly differentiated neuroendocrine histology tumor histologies with high prevalence of DLL3 (≥50% prevalence of ≥1% positivity), including but not limited to: melanoma, medullary thyroid cancer, esthesioneuroblastoma, bladder cancer, testicular cancer, glioblastoma multiforme, cervical cancer; large cell neuroendocrine tumor of lung, non-small cell lung cancers with mixed neuroendocrine features, and Merkel cell carcinoma OR
   4. DLL3+ (≥1% by IHC) Note: If patients are DLL3 negative per IHC but have a DLL3 prevelant tumor type, they will be allowed to enroll on the study.
4. Subjects who progressed or recurred after at least one line of therapy and are considered treatment refractory per standard of care.
5. Subjects willing to provide archived tumor tissue samples (formalin fixed, paraffin embedded [FFPE] sample). If no archived tumor tissue is available, we request to undergo pretreatment tumor biopsy. Subjects who do not have archived tumor tissue available and are unable or unwilling to undergo a pretreatment tumor biopsy due to extenuating circumstances (i.e., cannot be performed safely or inaccessible, as determined by the investigator) may be allowed to enroll without a tumor biopsy upon agreement with sponsor.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Minimum life expectancy of 12 weeks.
8. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
9. Measurable lesions as defined per RECIST 1.1 within 28 days prior to the first dose of tarlatamab.
10. Eligible for external beam radiation therapy to a previously unirradiated, measurable lesion as per standard of care.

    1. For the concurrent / sequential cohort of extracranial RT sites:

    i. A minimum of 10 subjects with thoracic lesions (lung, mediastinum, thoracic spine, rib, or other thoracic sites) will be treated ii. Subjects with treated brain metastases are eligible (untreated brain metastases are ineligible) provided they meet the following criteria:

<!-- -->

1. Definitive therapy was completed at least 2 weeks prior to the first dose of tarlatamab.
2. There is no evidence of radiographic central nervous system (CNS) progression following therapy and by the time of study screening.
3. Patients manifesting progression in lesions previously treated with stereotactic radiosurgery may still be eligible if pseudoprogression can be demonstrated by appropriate means.
4. Any CNS disease is asymptomatic for at least 7 days (unless symptoms are deemed irreversible by the investigator), the patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the subject is off or on stable doses of anti-epileptic drugs for malignant CNS disease for at least 7 days.

   b. For the concurrent/sequential cohort of cranial RT sites: i. Previously untreated brain lesions / metastases are eligible ii. Subjects with previously irradiated brain lesions are eligible provided they meet one of the following criteria:

<!-- -->

1. Prior PCI or whole brain radiation therapy per standard of care with new and/or recurrent brain metastases to be treated with SRS or hfSRT
2. Prior course(s) of SRS or hfSRT or other localized therapy with new lesion(s) to be treated with whole brain radiation therapy iii. Whole brain re-irradiation will be ineligible iv. Re-irradiation with SRS or hfSRT of previously irradiated lesion with SRS or hfSRT will be ineligible v. Craniospinal irradiation will not be allowed c. For the tarlatamab monotherapy cohort: i. Patient must have at least one measurable lesion, however that lesion does not need to be amenable to RT

1. Patients with previously irradiated lesions that have recurred or progressed are eligible 11. Adequate organ function, defined as follows:

a. Hematological function: i. Absolute neutrophil count ≥ 1.5 x 109/L ii. Platelet count ≥ 100 x 109/L iii. Hemoglobin > 9 g/dL (90 g/L) b. Coagulation function: i. Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 x institutional upper limit of normal (ULN). Subjects on chronic anticoagulation therapy who do not meet the criteria above may be eligible to enroll after discussion with the medical monitor.

c. Renal function: i. Estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) calculation > 30 mL/min/1.73 m2 d. hepatic function: i. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) < 3 x ULN (or < 5 x ULN for subjects with liver involvement) ii. Total bilirubin < 1.5 x ULN (or < 2 x ULN for subjects with liver metastases) e. Pulmonary function: i. No clinically significant pleural effusion ii. Baseline oxygen saturation > 90% on room air f. cardiac function (if obtained as part of standard of care): i. Cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and no clinically significant electrocardiogram (ECG) findings

Exclusion Criteria:

Re-irradiation, unless it is SRS/hfSRT after whole-brain radiation therapy (WBRT) or PCI or WBRT after SRS/hfSRT; re-irradiation of same lesion, unless verified with the Principal Investigator; patients with lesions not amenable to RT (including previously irradiated) will be only allowable on the tarlatamab monotherapy cohort.

Disease Related

1. Subjects are excluded from the study if any of the following criteria apply:

   1. No lesion(s)/site(s) amenable to radiation therapy (only eligible for tarlatamab monotherapy if open)
   2. Planned re-irradiation of a previously irradiated site
   3. Leptomeningeal disease requiring craniospinal irradiation
2. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
3. Subjects who experienced recurrent pneumonitis (grade 2 or higher) or severe, life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.
4. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1, or to levels dictated in the eligibility criteria with the exception of alopecia or toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present and stable for > 21 days) which may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and Amgen.

Other Medical Conditions

1. Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of tarlatamab.
2. History of arterial thrombosis (i.e., stroke or transient ischemic attack) within 12 months of first dose of tarlatamab.
3. Subject with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of tarlatamab.

   NOTE: Simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment. Subjects requiring oral antibiotics who have been afebrile > 24 hours, have no leukocytosis and have no clinical signs of infection are eligible. Subjects who meet these criteria and who were previously on IV antimicrobials should have been off IV antimicrobials for > 48 hours.
4. History of hypophysitis or pituitary dysfunction.
5. Exclusion of hepatitis infection based on the following results and/or criteria:

   a. Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B).

   b. Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.

   c. Positive hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
6. Major surgery requiring hospitalization for more than 3 days within 28 days of first dose of tarlatamab.
7. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
8. Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
9. Human immunodeficiency virus (HIV) infection.

   1. Subjects with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines.

Prior/Concomitant Therapy

1. Subject received prior therapy with tarlatamab.
2. Prior anti-cancer therapy within 30 days prior to first dose of tarlatamab.

   Exceptions:

   a. Subjects who received conventional chemotherapy are eligible if at least 14 days have elapsed and if all treatment-related toxicity has been resolved to grade ≤ 1.
3. Has a diagnosis of immunodeficiency (i.e., positive/non-negative test for human immunodeficiency virus) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab.
4. The following vaccines (live and live-attenuated vaccines) are excluded during the following study periods:

   1. Screening and during study treatment: Live and live-attenuated vaccines are prohibited within 28 days prior to the first dose of tarlatamab and for the duration of the study.
   2. Live viral non-replicating vaccine (i.e., Jynneos) for Monkeypox infection is allowed during the study (except during cycle 1) in accordance with local standard of care (SOC) and institutional guidelines.
   3. End of study treatment: Live and live-attenuated vaccines can be used when at least 60 days (5 x half-life of tarlatamab) have passed after the last dose of tarlatamab.

Other Exclusions

1. Female subjects of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of tarlatamab. Contraception methods for female subjects include:

1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, and implantable)
3. Intrauterine device
4. Intrauterine hormonal-releasing system
5. Bilateral tubal ligation/occlusion
6. Vasectomized partner (provided that partner is the sole sexual partner of the female subject of childbearing potential and that the vasectomized partner has received medical assessment of the surgical success)
7. Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments; the reliability of sexual abstinence must be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the subject) 2. Female subjects who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab.

   3. Female subjects planning to become pregnant while on study through 60 days after the last dose of tarlatamab.

   4. Female subjects of childbearing potential with a positive pregnancy test assessed at screening and/or day 1 by a highly sensitive urine or serum pregnancy test.

   5. Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception (use a condom) during treatment and for an additional 60 days after the last dose of tarlatamab.

   6. Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab.

   7. Male subjects unwilling to abstain from donating sperm during treatment and for an 60 days after the last dose of tarlatamab.

   8. Subject has known sensitivity to any of the products or components to be administered during dosing.

   9. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (i.e., Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.

   10. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing dose limiting toxicities (DLT) attributed to radiation or combination of radiation and tarlatamab. | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  The primary endpoint is safety, which will be measured by DLT using adverse events graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0) and ASTCT (CRS and ICANS). DLT will be defined as having 1) grade 3 - 5 non-hematologic adverse events (AEs) possibly, probably or definitely related to protocol treatment (radiation or combination of radiation and tarlatamab) by 8 weeks from start of radiation therapy; or 2) AEs possibly, probably, or definitely related to radiation or combination of radiation and tarlatamab leading to early termination of radiation or permanent discontinuation of tarlatamab. Grade 3+ AEs (or discontinuation) due to tarlatamab alone (not attributable to combination therapy) will not contribute to the primary endpoint. Frequency (%) of the patients with DLT will be reported by cohort.

SECONDARY OUTCOMES:
Objective response rate (ORR) using RESIST/iRECIST and RANO/RANO-BM criteria of radiated and non-radiated sites stratified by anatomic RT site and tumor histology. | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  ORR is defined as the percentage of subjects with measurable disease who have at least 1 confirmed response of complete response (CR) or partial response (PR) prior to any evidence of progression. ORR will be reported by cohort and site.
Toxicity of tarlatamab in tumors in all patients, not of SCLC histology, and stratified by histology in accordance with CTCAE v5. | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  Assess toxicity of therapy (tarlatamab with radiation therapy) by the incidence of treatment emergent adverse events reported (to include SAEs and AEs leading to discontinuation) based on CTCAE v5 and ASTCT (CRS and ICANS), stratified by histology and by SCLC vs. tumors that are not SCLC. Counts of all AEs by grade will be provided by cohort.
Overall survival (OS) | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  OS is defined as the time from registration to death and will be estimated using the Kaplan Meier method by cohort.
Progression free survival (PFS) | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  PFS according to RECIST guidelines is defined as the time from registration to progressive disease or death, whichever occurs first, and will be estimated using the Kaplan Meier method by cohort and site if applicable.
Duration or Response (DOR) | Until radiographic or disease progression or up to 24 months, whichever is earlier.
  DOR will only be evaluated in participants with objective response of CR or PR. All confirmed responders will be followed for at least 6 months from the onset of initial response. The end of response will match with the date of progression or death from any cause used for the PFS endpoint. The DOR estimate will be summarized using Kaplan-Meier method by cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hsu, MD, Principal Investigator — University of Arizona; Ricklie Julian, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at UMC North/University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No